CLINICAL TRIAL: NCT02569684
Title: Effects of Prebiotics on GLP-1 in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Diabetes Association (Other); Norwegian Extra Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, Anne-Marie Aas, Associate professor, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1180 REK
Record Dates: First submitted 2015-09-29; First posted 2015-10-07 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Inulin; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm A (Active Comparator): Prebiotic fibers: Oligofructose and inulin
  Interventions: Dietary Supplement: Prebiotic fibers: oligofructose and inulin
- Arm B (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Prebiotic fibers: oligofructose and inulin
  Arms: Arm A
Dietary Supplement: Maltodextrin
  Arms: Arm B

SUMMARY:
The aim of the study is to compare the effects of prebiotics versus placebo on blood concentrations of glucagon-like peptide-1 in subjects with diabetes type 2.

DETAILED DESCRIPTION:
We looked at 6 weeks supplementation with a prebiotic fibre mix of inulin and FOS. Cross over design compared to maltodextrin as placebo. Additional outcome measures: blood glucose, insulin, GLP-2, ghrelin, PYY and leptin after a standardized mixed meal test. Also measured changes in microbiota composition and SCFA in feces before and after intervention/placebo periods, and subjective measures of appetite.

ELIGIBILITY:
Inclusion Criteria:

* diabetes type 2
* BMI 18,5 - 40
* Not medicated with insulin, GLP-1 analogues or DPP4 inhibitors
* Moderate intake of alcohol
* Not excessive exercise
* Less than 3 kg weight change the last two months
* Intake of less than 30 g dietary fiber per day

Exclusion Criteria:

* IBD
* IBS
* Coeliac disease
* Have used antibiotics within the last two months
* Have used supplements with prebiotics or probiotics the last two months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Changes in plasma GLP-1 in response to standardized test meal before and after six weeks of ingestion of prebiotic fibers or placebo | six weeks
  The changes in GLP-1 response to either prebiotic fibers or placebo will be compared in a cross-over manner where the participants are their own controls. In between the intervention periods there will be a wash-out period of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Aas, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birkeland E, Bamigbetan WA, Molven KD, Thorsby PM, Gulseth HL, Aas AM, Dahl C. Can supplements with prebiotic fibres positively influence bone health in type 2 diabetes? Insights from a randomised controlled crossover trial. Arch Osteoporos. 2025 Jun 5;20(1):71. doi: 10.1007/s11657-025-01556-x. PMID 40471453
- [Derived] Birkeland E, Gharagozlian S, Gulseth HL, Birkeland KI, Hartmann B, Holst JJ, Holst R, Aas AM. Effects of prebiotics on postprandial GLP-1, GLP-2 and glucose regulation in patients with type 2 diabetes: A randomised, double-blind, placebo-controlled crossover trial. Diabet Med. 2021 Oct;38(10):e14657. doi: 10.1111/dme.14657. Epub 2021 Aug 7. PMID 34297363
- [Derived] Birkeland E, Gharagozlian S, Birkeland KI, Valeur J, Mage I, Rud I, Aas AM. Prebiotic effect of inulin-type fructans on faecal microbiota and short-chain fatty acids in type 2 diabetes: a randomised controlled trial. Eur J Nutr. 2020 Oct;59(7):3325-3338. doi: 10.1007/s00394-020-02282-5. Epub 2020 May 21. PMID 32440730